CLINICAL TRIAL: NCT06502444
Title: Moving Forward Together 2.0: An Activity Intervention
Acronym: MFT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: An insufficient number of prospective volunteers provided informed consent to provide a fair test of whether the intervention would be effective. More people were needed to make shared online feedback and support a useful component.
Sponsor: Rosalind Franklin University of Medicine and Science (Other)
Responsible Party: Principal Investigator, David Kosson, Professor, retired, Rosalind Franklin University of Medicine and Science
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHP23-428
Record Dates: First submitted 2024-06-14; First posted 2024-07-16 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Activity, Motor; Emotion Regulation
Keywords: activity; activity intervention; Post-traumatic Stress Disorder; intimate partner violence
MeSH Terms: conditions — Motor Activity; Emotional Regulation; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: The proposed design is a single condition, longitudinal pilot study examining the feasibility of using an online physical activity program to increase physical activity and improve emotion regulation in women who have experienced trauma due to experiencing an abusive or harmful relationship.
Masking Description: There is only one condition. All participants know they are signing up for this one condition, an activity intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Moving Forward Together Activity Intervention (Experimental): This is a single-arm project. All participants receive the same experimental intervention. The intervention is a gentle program encouraging greater participation in physical activity and healthy regulation of emotions.
  Interventions: Behavioral: Moving Forward Together Activity Intervention

INTERVENTIONS:
Behavioral: Moving Forward Together Activity Intervention — The activity intervention program consists of videos and handouts to encourage participants to access these materials if they wish to increase their physical activity. The program lasts 8 weeks. Participants may access program materials for an additional four weeks after the program ends

SUMMARY:
The study will test whether an online physical activity program that includes mindfulness can increase activity in women who have been abused by a relationship partner. The study also aims to test whether this intervention can improve their ability to control their emotions and use mindfulness and reduce their stress and Post-Traumatic Stress Disorder (PTSD) symptoms. The intervention is on the internet and provides participants with informational videos, as well as support and encouragement from other program participants. The intervention aims to encourage participants to choose their own physical activities and also includes components designed to foster healthy regulation of emotion (addressing negative thoughts and feelings that may get in the way of exercise, recognizing accomplishments and rewarding oneself, etc.) This activity intervention is designed to take eight weeks. Participants are tested initially (at baseline), halfway through the program (Week 4) and at the end of the program (Week 8).

DETAILED DESCRIPTION:
The proposed design is a single condition, longitudinal pilot study examining the feasibility of using an online physical activity program to increase physical activity and improve emotion regulation in women who have experienced trauma due to experiencing an abusive or harmful relationship. All participants receive the same intervention. The study will be conducted on the online Wix Classroom platform, which is a secure, online platform to which only participants and research staff will have access. Women who have varying levels of trauma, as determined by the PTSD Checklist-Civilian (PCL-C), will be invited to participate in the study via A Safe Place, an organization to help survivors of intimate partner violence. Participants will complete the online program, and are asked to complete assessments at baseline, 4 weeks, and 8 weeks. Though they will not be required to access the program, their continued use of the program after the end of the 8-week program will be examined for 4 additional weeks. The primary aim of this study is to assess the feasibility of the intervention. Descriptive statistics will be conducted to assess participant engagement (i.e., number of logins, video views, and discussion board posts) and satisfaction (i.e., program acceptability questionnaire responses). Feasibility data will help discern what program components participants found most useful. Longitudinal models will be used to examine the effect of program participation on physical activity, mood and emotion regulation, stress levels, and PTSD symptoms over time.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Female
* Reporting a previous relationship with an individual that included abuse or trauma
* Capable of reading and understanding English
* Not currently living with the individua
* Currently involved with A Safe Place in Zion, IL

Exclusion Criteria:

* Women without reliable internet access
* Individuals already meeting physical activity guidelines (150 minutes of physical activity or more per week)
* Women who report health problems that make activity unsafe or for whom healthcare professionals believe activity might be unsafe

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — women
Enrollment: 0 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Global Physical Activity Questionnaire | This measure is completed at baseline and at the eight-week assessment
  A 16-item measure of physical activity participation / sedentary behavior across three settings. We will assess whether participants engage in 150 minutes or more of leisure time physical activity per week. Those who do are ineligible for this study.
Post-traumatic Stress Disorder Checklist-Civilian (PCL-C): | This measure is completed at baseline and at the 4-week and 8-week assessment
  The PCL-C is a 17-item validated measure used to assess the intensity and severity of symptoms of Post-Traumatic Stress Disorder (PTSD). Each of the items is scored 1 to 5, so scores range from 17 to 85; higher scores indicate more symptoms of PTSD.
Positive and Negative Affect Schedule (PANAS) | This measure is completed at baseline and at the 8-week assessment
  The PANAS is a 20-item method for assessing both positive and negative affect. The Positive and Negative Affect Scales contain ten items each. Items are scored 1 to 5, so total subscale scores range from 10 to 50, where higher scores indicate greater levels of positive or negative emotion.
Emotion Regulation Questionnaire (ERQ) | This measure is completed at baseline, at the 4-week, and at the 8-week assessment.
  The ERQ is a 10-item measure used to assess participants' habitual use of two emotion regulation strategies: cognitive reappraisal (5 items) and expressive suppression (5 items). Scores on each item range from 1 to 7, so the range of subscale scores is 5 to 35, where higher scores indicate greater reliance on reappraisal or suppression.
Program acceptability measure. | This measure is only completed at the 8-week assessment.
  This 32-item measure assesses participants' experience of the online program. Participants also self-report their use of the different intervention components and the extent to which they found each component useful. There are 26 questions about participants' satisfaction with the program scored from 1 to 5. Scores will range from 1 to 150 where higher scores indicate greater satisfaction. There are also three questions about frequency of using different program features (scored from 0 to 6; range = 0 to 18; higher scores indicate greater frequency of using program elements. There is one question assessing the number of activity program units participants watched (ranging from 0 to 8, where a higher score indicates greater use of program material). There are 2 questions about participants' interest in continuing to access program materials. No scores will be computed from these questions.
Physical activity progress. | This measure is completed weekly for eight weeks
  Participants will be asked to share their physical activity tracking for each of the eight weeks of the program by reporting on their daily minutes of physical activity using a provided worksheet.
Affect Grid (Russell et al., 1989). | This measure is completed weekly for eight weeks
  This single item measure assesses both activation and valence associated with emotional response. Participants will be asked to report their current emotional state on a 9 X 9 grid that provides information about the valence of their emotional state (from extremeley unpleasant to extremely pleasant) and the intensity (or arousal) of their emotional state (from extreme sleepiness to extreme arousal). Participants' grid choices can be scored as self-ratings of affective valence and intensity on a scale that ranges from 1 to 9 in each case. In short, valence and intensity scores will range from 1 to 9 each week, where higher scores indicate more positive feelings and more intense feelings, respectively.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | This measure is completed at baseline, at the 4-week, and at the 8-week assessment.
  The 10-item Perceived Stress Scale assesses the level of stress partcipants perceive in their lives. Each item is scored 0 to 4, so total scores can range from 0 to 40, where higher scores indicate reports of greater perceived stress.
Online program use | Online program use is tracked separately for the eight-week program and for the four weeks following the end of the program
  Data from the online program will be extracted to track participants' use of the online program. Number of logins, number of video views, and number and content from discussion board posts will be extracted for each week of the online program, and during the 4 weeks the program website remains open after the 8-week program has ended

CONTACTS AND LOCATIONS:
Overall Officials: David Kosson, PhD, Principal Investigator — Rosalind Franklin University of Medicine and Science; Steven Miller, PhD, Principal Investigator — Rosalind Franklin University of Medicine and Science
Locations (2):
- United States (2):
  - Rosalind Franklin University of Medicine and Science, North Chicago, Illinois
  - A Safe Place, Zion, Illinois

IPD SHARING:
Plan to Share IPD: No
Data collected in this study will not be shared with researchers outside of the identified research personnel.

REFERENCES:
- [Background] Cohen S, Williamson, G. Perceived stress in a probability sample of the United States. In: Spacapan, S, Oskamp, S, ed. The social psychology of health: Claremont symposium on applied social psychology. Newbury Park, CA: Sage; 1988:31-57. www.cmu.edu/dietrich/psychology/stress-immunity-disease-lab/scales/pdf/cohen,-s.--williamson,-g.-1988.pdf
- [Background] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Bull FC, Maslin TS, Armstrong T. Global physical activity questionnaire (GPAQ): nine country reliability and validity study. J Phys Act Health. 2009 Nov;6(6):790-804. doi: 10.1123/jpah.6.6.790. PMID 20101923
- [Background] Neumann CS, Pardini D. Factor structure and construct validity of the Self-Report Psychopathy (SRP) scale and the Youth Psychopathic Traits Inventory (YPI) in young men. J Pers Disord. 2014 Jun;28(3):419-33. doi: 10.1521/pedi_2012_26_063. Epub 2012 Sep 17. PMID 22984856
- [Background] Karstoft KI, Andersen SB, Bertelsen M, Madsen T. Diagnostic accuracy of the posttraumatic stress disorder checklist-civilian version in a representative military sample. Psychol Assess. 2014 Mar;26(1):321-5. doi: 10.1037/a0034889. Epub 2013 Nov 4. PMID 24188155
- [Background] Russell JA, Weiss A, Mendelsohn, GA. Affect grid: A single item scale of pleasure and activation. J Pers Soc Psychol. 1989; 57, 493-502. http://dx.doi.org/10.1037/0022-3514.57.3.493